CLINICAL TRIAL: NCT05348733
Title: FINE-REAL: A Non-interventional Study Providing Insights Into the Use of Finerenone in a Routine Clinical Setting
Brief Title: A Study Called FINE-REAL to Learn More About the Use of the Drug Finerenone in a Routine Medical Care Setting
Status: Recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21785
Record Dates: First submitted 2022-04-01; First posted 2022-04-27 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2 | interventions — finerenone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants diagnosed with CKD and T2D: Participants who are newly prescribed finerenone under routine treatment conditions.
  Interventions: Drug: Kerendia (Finerenone, BAY94-8862)

INTERVENTIONS:
Drug: Kerendia (Finerenone, BAY94-8862) — Decision will taken by the treating physician to initiate treatment with finerenone.

SUMMARY:
This is an observational study in people with chronic kidney disease (CKD) and type 2 diabetes (T2D) who will be receiving finerenone.

Kidneys filter extra water and waste out of the blood and make urine. CKD is a long-term, progressive, decrease in the kidneys' ability to filter the blood properly. In people with T2D, the body does not make enough of a hormone called insulin, or does not use insulin well enough, resulting in high blood sugar levels that can cause damage to the kidneys. As a result, CKD can occur as a complication of T2D.

Finerenone works by blocking certain proteins, called mineralocorticoid receptors. An increased stimulation of these proteins is thought to damage the kidneys and the heart. By lowering their stimulation, finerenone reduces the risk of kidney disease progressively getting worse.

Finerenone is available and approved for doctors to prescribe to people with CKD and T2D. Since it has only recently become available for these patients, there is a need for more information about the use of finerenone in the real-world setting.

The main purpose of the study is to learn more about treatment patterns in people with CKD and T2D who just started or will start finerenone treatment as decided and prescribed by their doctor as part of their routine medical care.

To answer this question, the researchers will collect data on:

* Clinical characteristics (e.g., history of CKD and T2D, blood pressure, heart health) of the participants
* Reasons for starting finerenone
* Reasons for stopping finerenone early
* How long participants have been taking finerenone (planned by their doctor compared to actual time it was taken)
* Dosing of finerenone
* Other medications used while taking finerenone

The researchers will also collect data on medical problems (called adverse events) that the participants may have during the study. All adverse events are collected, even if they might not be related to the study treatment.

Hyperkalemia, a medical term used to describe a potassium level in the blood that is higher than normal, is of special interest when finerenone is combined with some medications commonly taken to control blood pressure. Researchers want to know how often higher potassium levels occur, and when it leads to:

* Stopping finerenone treatment too early
* Dialysis (a medical procedure to filter the blood of extra water and waste)
* Care in a hospital

All data will come from medical records or from interviews study doctors will have with the participants during visits that take place during routine medical care.

Participants in the US will be invited to provide voluntary blood and urine samples that could be analyzed later to better understand possible changes in protein or nucleic acid levels over time.

Each participant will be in the study for 12 months. This time participating in the study may be shorter if their finerenone treatment is stopped early or the study comes to an end as planned in September 2027.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants of all genders (≥18 years old)
* Diagnosis of CKD associated with T2D based on assessment by physician.
* Treatment according to local marketing authorization, finerenone 20 or 10 mg.Treatment should have been started up to 8 weeks before or after the ICF is signed.
* Decision to initiate treatment with finerenone must be made before ICF is signed.
* Signed informed consent

Exclusion Criteria:

* Participation in an investigational trial at any time during the course of this study
* Contra-indications according to the local label.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a diagnosed of CKD and T2D will be enrolled after the decision for treatment with finerenone has been made by the treating physician.
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Descriptive analysis of clinical characteristics of participants with chronic kidney disease (CKD) and with type 2 diabetes(T2D). | Approximately 62 months
Descriptive summary of reasons for introducing finerenone. | Approximately 62 months
Descriptive summary of reasons for discontinuation of finerenone. | Approximately 62 months
Planned and actual duration of treatment with finerenone | Approximately 62 months
Planned and actual daily dose of finerenone treatment | Approximately 62 months
Planned and actual frequency of finerenone treatment | Approximately 62 months
Descriptive summary of secondary therapies used in participants with CKD and T2D. | Approximately 62 months

SECONDARY OUTCOMES:
Occurrence of adverse events (AEs) and serious adverse events (SAEs) | Approximately 62 months
Occurrence of hyperkalemia | Approximately 62 months
  leading to permanent study drug discontinuation, dialysis or hospitalization

OTHER OUTCOMES:
Descriptive summary for healthcare resource utilization. | Approximately 62 months
Occurrence of newly diagnosed diabetic retinopathy or progression of existing disease at treatment initiation | Approximately 62 months

CONTACTS AND LOCATIONS:
Locations (68):
- United States (49):
  - Nephrology Consultants LLC, Huntsville, Alabama
  - AKDHC Medical Research Servies LLC, Phoenix, Arizona
  - Harrisburg Family Medical Center, Harrisburg, Arkansas
  - Kidney Disease Medical Group, Glendale, California
  - Renal Consultants Medical Group, Granada Hills, California
  - Keck School of Medicine of University of Southern California, Los Angeles, California
  - UCSF Nephrology Clinic, San Francisco, California
  - University of Central Florida College of Medicine, Orlando, Florida
  - Gulf View Medical, Port Charlotte, Florida
  - Hanson Clinical Research Center, Port Charlotte, Florida
  - Metabolic Research Institute, West Palm Beach, Florida
  - Ellipsis Group, Alpharetta, Georgia
  - Augusta University, Augusta, Georgia
  - Coastal Medical Research, Brunswick, Georgia
  - Caritas Medical Center, Stockbridge, Georgia
  - Herman Clinical Research LLC, Suwanee, Georgia
  - Laurie Tom, MD, Honolulu, Hawaii
  - Pacific Diabetes & Endocrine Center, Honolulu, Hawaii
  - Cook County Health, Chicago, Illinois
  - Jesse Brown VA Medical Center, Chicago, Illinois
  - Medico, Chicago, Illinois
  - Nephrology Associates Northern Illinois and Indiana, Hinsdale, Illinois
  - Kidney and Hypertension Center of Wabash Valley LLC, Terre Haute, Indiana
  - University of Iowa Preventive Intervention Clinic, Iowa City, Iowa
  - Northwest Louisiana Nephrology, Shreveport, Louisiana
  - Ochsner Medical Foundation, Slidell, Louisiana
  - University of Maryland Midtown Professionals Group Healthcare, Baltimore, Maryland
  - NECCR Primacare Research, LLC, Fall River, Massachusetts
  - Healthy Heart Cardiology, Grand Rapids, Michigan
  - Care Access Research - Minneapolis, Minneapolis, Minnesota
  - Jackson Medical Mall University Home Dialysis Clinic, Jackson, Mississippi
  - Nephrology and Hypertension Associates, Tupelo, Mississippi
  - Renown Regional Medical Center, Reno, Nevada
  - The EnLyv Clinics, Edison, New Jersey
  - Gaffney Health Services, Charlotte, North Carolina
  - Bland Clinic, Greensboro, North Carolina
  - Ardmore Medical Research, Winston-Salem, North Carolina
  - Panoramic Health, Providence, Rhode Island
  - DarSalud Care / LifeDOC Research, Memphis, Tennessee
  - Academy of Diabetes Thyroid and Endocrine, El Paso, Texas
  - AA Medical Research Center, Flint, Texas
  - Prolato Clinical Research, Houston, Texas
  - Clinical Research Stategies Inc, Houston, Texas
  - RGV Endocrine Center, McAllen, Texas
  - Dallas Renal Group, Plano, Texas
  - Tranquil Clinical Research, Webster, Texas
  - University of Utah, Salt Lake City, Utah
  - Washington Nephrology Associates, Alexandria, Virginia
  - MultiCare Endocrinology Specialists Tacoma, Tacoma, Washington
- Many Locations, Multiple Locations, Argentina
- Many Locations, Multiple Locations, Belgium
- Many Locations, Multiple Locations, Brazil
- Many Locations, Multiple Locations, Canada
- Many Locations, Multiple Locations, China
- Many Locations, Multiple Locations, Denmark
- Many Locations, Multiple Locations, Germany
- Many Locations, Multiple Locations, Greece
- Many Locations, Multiple Locations, Mexico
- Many Locations, Multiple Locations, Netherlands
- Many Locations, Multiple Locations, Portugal
- Many Locations, Multiple Locations, Russia
- Many Locations, Multiple Locations, Saudi Arabia
- Many Locations, Multiple Locations, Singapore
- Many Locations, Multiple Locations, Slovenia
- Many Locations, Multiple Locations, South Korea
- Many Locations, Multiple Locations, Switzerland
- Many Locations, Multiple Locations, Taiwan
- Many Locations, Multiple Locations, Thailand

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Mottl A, Scott C, Green JB, Heerspink HJL, Mann JFE, McGill JB, Nangaku M, Rosenstock J, Rossing P, Li L, Li N, Vaduganathan M, Agarwal R; CONFIDENCE Trial Investigators. Baseline Kidney Function, Albuminuria, and Urine Albumin-Creatinine Ratio Reduction with Finerenone, Empagliflozin, or Both: Post Hoc Analyses of CONFIDENCE Trial. J Am Soc Nephrol. 2025 Nov 6. doi: 10.1681/ASN.0000000928. Online ahead of print. No abstract available. PMID 41196655
- [Derived] Desai NR, Navaneethan SD, Nicholas SB, Pantalone KM, Wanner C, Hamacher S, Gay A, Wheeler DC. Design and rationale of FINE-REAL: A prospective study of finerenone in clinical practice. J Diabetes Complications. 2023 Apr;37(4):108411. doi: 10.1016/j.jdiacomp.2023.108411. Epub 2023 Feb 2. PMID 36857997
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — https://clinicaltrials.bayer.com